CLINICAL TRIAL: NCT01032902
Title: Study to Establish the Ability of the Chembio Diagnostics Systems, Inc. DPP HIV 1/2 Rapid Test to Qualitatively Detect the Presence of Antibodies Against HIV-1 in Oral Fluid, Whole Blood (Capillary and Venous), Serum and Plasma
Brief Title: Evaluation of the Performance of Chembio Diagnostics Systems, Inc. DPP® HIV 1/2 Rapid Test
Status: Completed | Type: Observational
Sponsor: Chembio Diagnostic Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-HIV01; IDE 14208
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: HIV Infections
Keywords: Human immunodeficiency virus; Rapid Test; HIV; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Reagent Kits, Diagnostic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Known HIV positive: Patients from HIV clinics with documented infections
  Interventions: Device: In Vitro Diagnostic Device
- High Risk for Infection with HIV: Patients from defined HIV high-risk populations - i.e. intravenous drug users, or patients presenting with symptoms of sexually transmitted disease.
  Interventions: Device: In Vitro Diagnostic Device
- Low-Risk for Infection with HIV: Individuals not known to belong to any of the defined high-risk groups - i.e. "healthy patients" presenting for routine physicals or other unrelated non-life threatening illnesses, or individuals from a general low risk population such as students, employees of academic or other institutions, etc…
  Interventions: Device: In Vitro Diagnostic Device

INTERVENTIONS:
Device: In Vitro Diagnostic Device — For the detection of antibodies to HIV in serum, plasma, blood and oral fluid

SUMMARY:
This study has been designed to evaluate the performance of the Chembio Diagnostics Systems, Inc. DPP® HIV 1/2 rapid test. The device is intended to qualitatively detect the presence of antibodies against HIV-1/2 in oral fluid, whole blood (capillary and venous), serum or plasma. This study will assess the DPP® HIV 1/2 Screen assay's ability to detect HIV-1.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 2 years of age (no upper age limit).
* Must be willing and able to receive post-test counseling, if applicable.
* Must sign (and be given) a copy of the written Informed Consent form and or Assent form (if applicable).
* Must be able to sustain fingersticks and venipuncture from the arm or hand only.

Exclusion Criteria:

* Am in a life threatening condition at the time of enrollment
* Have a suppressed immune systems (i.e. transplant patients, individuals diagnosed with non-HIV immunosuppressive illness, etc.).
* Have participated or are participating in a clinical trial for an HIV vaccine.
* Have previously participated in this clinical trial.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Point-of-care test sites including clinics and physician office settings
Sampling Method: Non-Probability Sample
Enrollment: 2808 (Actual)
Dates: Start 2010-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The device detects HIV-1 antibodies in a variety of sample matrices: capillary whole blood, venous whole blood (with EDTA or heparin anticoagulant), oral fluid, serum and plasma (with EDTA or heparin anticoagulant). | 20 minutes

SECONDARY OUTCOMES:
The device provides a qualitative screen for the detection of antibodies to HIV-1 compared to an FDA approved HIV-1/2 EIA, with sensitivity and specificity equal to or greater than 98% at the lower 95% confidence interval boundary. | 20 minutes

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Univeristy of California, San Diego, La Jolla, California
  - Therafirst, Fort Lauderdale, Florida
  - University of Maryland, Baltimore, Maryland
  - St. Christopher's Hospital for Children/ Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Texas HSC, Houston, Texas